CLINICAL TRIAL: NCT04185662
Title: Effects of Artificial Sweeteners on Glucose Metabolism in Patients With Type 2 Diabetes -A Multi-Center Randomized Controlled Clinical Trial(SWEETS)
Brief Title: Effects of Artificial Sweeteners on Glucose Metabolism in Patients With Type 2 Diabetes
Acronym: SWEETS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: ShiBei Hospital , JingAn District, Shanghai (Unknown); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); PuNan Hospital ,Shanghai (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: T2DM20190619
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: artificial sweetners; glucose metabolism; type 2 diabetic patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trichlorosucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- placebo (Placebo Comparator): intake 200 ml water daily for 3 months
  Interventions: Dietary Supplement: sucralose
- low dose sucrolose group (Experimental): intake 12.3mg sucralose in 200 ml water daily for 3 months
  Interventions: Dietary Supplement: sucralose
- moderate dose sucrolose group (Experimental): intake 73.8mg sucralose in 200ml water daily for 3 months
  Interventions: Dietary Supplement: sucralose

INTERVENTIONS:
Dietary Supplement: sucralose — daily intake different dose of artificial sweeteners sucralose or placebo

SUMMARY:
To investigate the effects of artificial sweeteners on glucose metabolism in newly diagnosed type 2 diabetic patients

DETAILED DESCRIPTION:
Artificial sweeteners are among the most widely used food additives worldwide. Artificial sweeteners consumption is considered safe and beneficial owing to their low caloric content. However, recent studies demonstrated that consumption of commonly used artificial sweeteners formulations drives the development of glucose intolerance in healthy human subjects. However,the effects of artificial sweeter on glucose metabolism in newly diagnosed type 2 diabetic patients remains unknown. Thus, different doses of sweeteners will be given to newly diagnosed type 2 diabetic patients to investigate the effects of artificial sweeteners on glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed type 2 diabetes, diagnosed by World Health Organization criteria, were recruited from outpatient of the Endocrinology Department in Shanghai Renji Hospital, Shanghai PuNan hospital，Shanghai ShiBei hospital, shanghai xinhua hospital, chongming branch;
* FBG≤ 9 mmol/L, HbA1c≤ 7% ;without any oral hypoglycemic agents or insulin,
* Age ≥30 and ≤ 60 years old.
* BMI >24 and <28 kg/m2; --no regular consumption of artificial sweeteners or foods that have added much sweeteners.(eg:Coca-Cola zero), no sucralose intolerance.

Exclusion Criteria:

* patients who had a history of acute and chronic diarrhea or constipation or severe chronic gastrointestinal disease..
* underwent enterectomy or other abdominal surgery (e.g., gallbladder removal) within one year;
* take antibiotics, antidiarrheic, antispasmodic, steroids and immune agents within three months.
* Patients who had a history of abnormal renal function(creatinine >132μmol/L), active liver disease(ALT were 2.5 times higher than the normal upper limit), or accompany with other sever diseases, such as severe infection, severe anemia, neutropenia and mental illness.
* Other serious heart disease, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated heart disease,cardiac function(NYHA) classification>level III.
* A history of acute complications such as diabetic ketoacidosis or hypertonic coma within 3 months.
* pregancy
* Allergic to sweeteners.
* participant in any clinical trail within 3 months

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose | 3 month
  Fasting glucose change from baseline
postprandial blood sugar | 3 month
  postprandial blood glucose change from baseline
HbA1c | 3 month
  HbA1c change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, professor, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No